CLINICAL TRIAL: NCT07023900
Title: Transvenous Lead Removal Only With Manual Traction Without Extraction Tools
Brief Title: Lead Extraction With Manual Traction
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Prof. Dr., Bursa Postgraduate Hospital
Other Study IDs: BursaPH Lead
Record Dates: First submitted 2025-06-01; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pacemaker Lead Dysfunction; Manual Traction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Manual traction — The pacemaker or ICD lead extraction with manually.

SUMMARY:
The number of implantable cardiac rhythm devices is increasing. As a result, the number of patients requiring lead extraction is increasing. In this study, authors aimed to present their experience with lead extraction using manual traction.

DETAILED DESCRIPTION:
Objectives: The number of implantable cardiac rhythm devices is increasing. As a result, the number of patients requiring lead extraction is increasing. In this study, authors aimed to present our experience with lead extraction using manual traction.

Methods: Patients (n=130) who underwent lead extraction by manual traction without the use of lead extraction devices (extraction sheaths, locking stylets, etc.) manufactured for extraction at our hospital between 2016 and 2021 were reviewed. Patient characteristics, indications for extraction, procedural success, complications, and mortality were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who underwent transvenous lead extraction manually
* Patients, who had lead and device types

Exclusion Criteria:

* Patients, who underwent transvenous lead extraction with extraction device
* Patients, who had not baseline characteristics
* Patients, who had not procedure detail

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent transvenous lead extraction manually in our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Extraction the pacemaker or ICD lead manually without complication. | one month
  The patients number of extraction of all lead and pacemaker generator components without major complications was defined as procedural success.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kusumoto FM, Schoenfeld MH, Wilkoff BL, Berul CI, Birgersdotter-Green UM, Carrillo R, Cha YM, Clancy J, Deharo JC, Ellenbogen KA, Exner D, Hussein AA, Kennergren C, Krahn A, Lee R, Love CJ, Madden RA, Mazzetti HA, Moore JC, Parsonnet J, Patton KK, Rozner MA, Selzman KA, Shoda M, Srivathsan K, Strathmore NF, Swerdlow CD, Tompkins C, Wazni O. 2017 HRS expert consensus statement on cardiovascular implantable electronic device lead management and extraction. Heart Rhythm. 2017 Dec;14(12):e503-e551. doi: 10.1016/j.hrthm.2017.09.001. Epub 2017 Sep 15. No abstract available. PMID 28919379
- [Background] Bongiorni MG, Burri H, Deharo JC, Starck C, Kennergren C, Saghy L, Rao A, Tascini C, Lever N, Kutarski A, Fernandez Lozano I, Strathmore N, Costa R, Epstein L, Love C, Blomstrom-Lundqvist C; ESC Scientific Document Group. 2018 EHRA expert consensus statement on lead extraction: recommendations on definitions, endpoints, research trial design, and data collection requirements for clinical scientific studies and registries: endorsed by APHRS/HRS/LAHRS. Europace. 2018 Jul 1;20(7):1217. doi: 10.1093/europace/euy050. No abstract available. PMID 29566158